CLINICAL TRIAL: NCT00416832
Title: Optimising Therapy for Boys With Hodgkin's Lymphoma and Quality Assurance of Therapy for Girls With Hodgkin's Lymphoma Until Start of a New Prospective Trial for Hodgkin's Lymphoma in Childhood and Adolescence
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Young Patients With Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christine Mauz-Körholz (Other)
Responsible Party: Sponsor-Investigator, Christine Mauz-Körholz, Prof. Dr. Christine Mauz-Körholz, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Purpose: Treatment
Other Study IDs: CDR0000514355; GPOH-HD-2002; EU-20651
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma
Keywords: stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Cyclophosphamide; Dacarbazine; Doxorubicin; Etoposide; Prednisone; Procarbazine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cyclophosphamide
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: prednisone
Drug: procarbazine hydrochloride
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill cancer cells. Giving combination chemotherapy together with radiation therapy may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects and how well giving combination chemotherapy together with radiation therapy works in treating young patients with Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of intensified etoposide administered as a part of OEPA combination chemotherapy (vincristine, etoposide, prednisone, and doxorubicin hydrochloride) in pediatric male patients with intermediate or advanced Hodgkin's lymphoma (HL).
* Determine the safety and efficacy of COPDIC combination chemotherapy (cyclophosphamide, vincristine, prednisone, and dacarbazine) or COPP combination chemotherapy (cyclophosphamide, vincristine, procarbazine hydrochloride, and prednisone) in reducing gonadotoxicity in male or female patients.
* Assess quality assurance of these regimens in pediatric female patients with intermediate or advanced HL.

OUTLINE: This is a pilot, multicenter study. Patients are stratified according to disease stage (I or IIA vs IIB, IIE, or IIIA vs IIBE, IIIBE, or IV).

* Stratum 1 (stages I or IIA): Male patients receive vincristine IV on days 1, 8, and 15, etoposide IV over 2 hours on days 3-7, oral prednisone on days 1-15, and doxorubicin hydrochloride IV over 4 hours on days 1 and 15 (OEPA). Female patients receive vincristine, prednisone, and doxorubicin hydrochloride as in male patients and oral procarbazine hydrochloride on days 1-15 (OPPA). Both regimens repeat every 4 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients who do not achieve complete remission undergo involved-field radiotherapy beginning 3 weeks after completion of chemotherapy.
* Stratum 2 (stages IIB, IIE, or IIIA): Male patients receive 2 courses of OEPA as in stratum 1 followed by 2 courses of COPDIC comprising oral prednisone on days 1-15, dacarbazine IV over 30 minutes on days 1-3, and vincristine IV and cyclophosphamide IV over 1 hour on days 1 and 8. Female patients receive 2 courses of OPPA as in stratum 1 followed by COPP comprising oral prednisone and 2 courses of oral procarbazine hydrochloride on days 1-15 and vincristine IV and cyclophosphamide IV over 1 hour on days 1 and 8. Both regimens repeat every 4 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning 3 weeks after completion of chemotherapy, all patients undergo involved-field radiotherapy.
* Stratum 3 (stages IIBE, IIIBE, or IV): Male patients receive 2 courses of OEPA as in stratum 1 followed by 4 courses of COPDIC as in stratum 2. Female patients receive 2 courses of OPPA as in stratum 1 followed by 4 courses of COPP as in stratum 2. Beginning 3 weeks after completion of chemotherapy, all patients undergo involved-field radiotherapy.

PROJECTED ACCRUAL: A total of 648 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of classic Hodgkin's lymphoma (HL)

  * Intermediate or advanced disease, including the following stages:

    * Stage I
    * Stage IIA, IIB, IIE, or IIBE
    * Stage IIIA or IIIBE
    * Stage IV

PATIENT CHARACTERISTICS:

* No other concurrent malignancies
* No severe concurrent diseases (e.g., immune deficiency syndrome)

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* Pre-phase therapy for large mediastinal tumor allowed

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 648 (Estimated)
Dates: Start 2002-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy
Reduction of gonadotoxicity
Quality assurance

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koerholz, MD, Study Chair — Martin-Luther-Universität Halle-Wittenberg